CLINICAL TRIAL: NCT04104763
Title: Osteofibrous Dysplasia (Kempson-Campanacci's Disease): Long Term Follow-up Study on Natural History, Results of Treatment and Relationship With Adamantinoma
Brief Title: Osteofibrous Dysplasia (Kempson-Campanacci's Disease)
Acronym: DOFOL
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Alberto Righi, Principal Investigator, Istituto Ortopedico Rizzoli
Other Study IDs: 9261_2019
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2021-08

CONDITIONS: Osteofibrous Dysplasia
MeSH Terms: conditions — Osteofibrous Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: study of osteofibrous dysplasia features — obtain long term follow-up in patients with osteofibrous dysplasia, to assess natural history of the disease, late results of treatment and in particular the potential and risk of progression to adamantinoma.

SUMMARY:
The aim of the present study is to obtain long term follow-up in patients with osteofibrous dysplasia, to assess natural history of the disease, late results of treatment and in particular the potential and risk of progression to adamantinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients treated at Rizzoli Institute from 01 Jan 1943 to 31 Dic 2011
* Diagnosis of osteofibrous dysplasia pathologically confirmed
* Written informed consent prior to any study-specific analysis and/or data collection

Exclusion Criteria:

* Patients with histological diagnosis different from osteofibrous dysplasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is single institution cases series review of histological and clinical data
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Osteofibrous Dysplasia (Kempson-Campanacci's disease): Long Term Follow-up Study on Natural History, Results of Treatment and Relationship with Adamantinoma | BASELINE
  We will retrieve from the database of the Rizzoli institute all the cases with a histological diagnosis of Ewing sarcoma from 01 Jan 1943 to 31 Dic 2011.
  We aspect to find approximately 55 cases. We will review all the medical records, radiological imaging, and histological data of these cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Pathology of IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Result] Benassi MS, Campanacci L, Gamberi G, Ferrari C, Picci P, Sangiorgi L, Campanacci M. Cytokeratin expression and distribution in adamantinoma of the long bones and osteofibrous dysplasia of tibia and fibula. An immunohistochemical study correlated to histogenesis. Histopathology. 1994 Jul;25(1):71-6. doi: 10.1111/j.1365-2559.1994.tb00600.x. PMID 7525449
- [Result] Scholfield DW, Sadozai Z, Ghali C, Sumathi V, Douis H, Gaston L, Grimer RJ, Jeys L. Does osteofibrous dysplasia progress to adamantinoma and how should they be treated? Bone Joint J. 2017 Mar;99-B(3):409-416. doi: 10.1302/0301-620X.99B3.38050. PMID 28249983
- [Result] Gleason BC, Liegl-Atzwanger B, Kozakewich HP, Connolly S, Gebhardt MC, Fletcher JA, Perez-Atayde AR. Osteofibrous dysplasia and adamantinoma in children and adolescents: a clinicopathologic reappraisal. Am J Surg Pathol. 2008 Mar;32(3):363-76. doi: 10.1097/PAS.0b013e318150d53e. PMID 18300815

DOCUMENTS (1):
  • Study Protocol (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT04104763/Prot_000.pdf